CLINICAL TRIAL: NCT00219921
Title: Postoperative Analgesia After Total Hip Replacement
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LTC-349-030905
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2007-03-30 (Estimated); Status verified 2007-03

CONDITIONS: Total Hip Replacement
Keywords: total hip replacement; pain treatment
MeSH Terms: conditions — Agnosia | interventions — Analgesia, Patient-Controlled; Morphine

INTERVENTIONS:
Drug: Intrathecal morphine at surgery, 0.1mg and placebo
Drug: Patient Controlled Analgesia with iv morphine and placebo
Drug: intrathecal morphine AND patient controlled analgesia with iv morphine

SUMMARY:
There are several treatments for postoperative pain after Hip Replacement Surgery. However, some require an intravenous line which may interfere with rehabilitation after surgery. This study aims to evaluate which method of pain treatment is best after Hip Replacement Surgery. Patients will either receive pain treatment at surgery, continuous intravenous pain treatment, or both. In the first two days after surgery, patients will frequently be asked to rate their pain, and use of other pain medication will be monitored.

DETAILED DESCRIPTION:
This is a three-group randomized placebo-controlled double blind trial to assess which postoperative analgesia is best after total hip replacement. The conventional analgesia includes both intrathecal morphine at surgery and Patient Controlled Analgesia (PCA) with morphine in the first 48 hours after surgery. This will be compared with two experimental groups which will receive either intrathecal morphine and PCA with placebo or intrathecal placebo and PCA with morphine. Escape medication with intramuscular morphine is available in all groups. A total of 120 patients will be randomized.

VAS- score at rest and with movement will be recorded every three hours for the first 48 hours after surgery, as well as PCA-bolussum and Morphine IM.

ELIGIBILITY:
Inclusion Criteria:

* Patients accepted for fast-track total hip replacement, i.e.ASA 3 or lower

Exclusion Criteria:

* Not able to speak dutch
* communication problems
* dementia
* mental retardation

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2005-09; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
VAS-score for pain at movement and at rest every three hours
PCA-bolus-sum every three-hour period
Morphine-IM rescue dose every three-hour period

SECONDARY OUTCOMES:
patient satisfaction each 24 hours
iv-morphine dose needed to attain VAS-score under 40 mm
PONV every three hours
urine retention every three hours
itching every three hours
decrease in saturation every three hours
quality of physical training

CONTACTS AND LOCATIONS:
Overall Officials: Sibrand Houtman, MD, Principal Investigator — Rijnstate Hospital